CLINICAL TRIAL: NCT06181539
Title: Evaluate the Effect of Prone Ventilation on Ventilated-blood Flow Ratio in Patients With Acute Respiratory Distress Syndrome by Electrical Impedance Tomography
Brief Title: Evaluate the Effect of Prone Ventilation on Ventilated-blood Flow Ratio in Patients With ARDS by EIT
Status: Completed | Type: Observational
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Sponsor
Other Study IDs: PPVEIT20230502
Record Dates: First submitted 2023-12-13; First posted 2023-12-26 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Acute Respiratory Distress Syndrome; Electrical Impedance Tomography; Prone Position Ventilation; Ventilation Perfusion Mismatch
Keywords: Acute Respiratory Distress Syndrome; Electrical impedance tomography; prone position ventilation
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Patients with ARDS often suffer a gravity-dependent alveolar collapse, resulting in a reduction of tidal volume, residual alveolar excessive distension, and ventilator-related lung injury(VILI) induced by unreasonable ventilator setting.Prone ventilation (PPV) improves the gravity-dependent alveolar ventilation and promotes lung recruitment in the gravity-dependent area and improves lung compliance. Previous studies showed that prolonged PPV combined with low tidal volume(LTV) lung protected ventilation can significantly reduce the mortality of patients with moderate to severe ARDS.Although more than 60% of patients with moderate to severe ARDS due to COVID-19 has been widely implemented PPV,studies showed an improvement in oxygenation in patients with ARDS(the P/F radio improved by more than 20% before and after PPV) was 9-77%, that is, That is, some patients are unresponsive to PPV. In addition, some patients showed CO2 responsiveness after PPV(ventilation rate (VR) decreased significantly after PPV).The tools for monitoring the effects of PPV on ventilation and blood flow at bedside are still lacking, Electrical impedance tomography (EIT) is a non-invasive, non-radiative, real-time bedside lung imaging technique that can monitor local lung ventilation distribution. This study intends to use EIT to evaluate pulmonary ventilation, blood flow distribution and local V/Q ratio before and after PPV, as well as to monitor the changes in pulmonary physiology before and after PPV, explore the mechanism of PPV improving oxygenation by combined with the changes in oxygenation, and explore the factors that predict and affect PPV responsiveness.

DETAILED DESCRIPTION:
Acute respiratory distress syndrome (ARDS) is presented as acute hypoxemia and pulmonary edema due to the increased permeability of alveolar capillaries. Endothelial damage injury and swelling, microthrombosis, and hypoxic pulmonary vasoconstriction can lead to low pulmonary blood vessels perfusion and even occlusion, while patients with ARDS often suffer a gravity-dependent alveolar collapse, resulting in a reduction of tidal volume, residual alveolar excessive distension, and ventilator-related lung injury(VILI) induced by unreasonable ventilator setting.Prone ventilation (PPV) improves the gravity-dependent alveolar ventilation and promotes lung recruitment in the gravity-dependent area and improves lung compliance. Besides, pulmonary blood perfusion is less affected by gravity distribution, thus the improvement of gravity-dependent alveolar ventilation can significantly reduce shunt, and lung heterogeneity and improve V/Q radio. Previous studies showed that prolonged PPV combined with low tidal volume lung protected ventilation can significantly reduce the mortality of patients with moderate to severe ARDS.Although more than 60% of patients with moderate to severe ARDS due to COVID-19 has been widely implemented PPV,studies showed an improvement in oxygenation in patients with ARDS(the P/F radio improved by more than 20% before and after PPV) was 9-77%, that is, That is, some patients are unresponsive to PPV. In addition, some patients showed CO2 responsiveness after PPV (ventilation rate (VR) decreased significantly after PPV).The tools for monitoring the effects of PPV on ventilation and blood flow at bedside are still lacking, Electrical impedance tomography (EIT) is a non-invasive, non-radiative, real-time bedside lung imaging technique that can monitor local lung ventilation distribution. By injecting hypertonic saline through a central vein catheter, we can obtain lung perfusion images to indicate local lung blood flow distribution. In addition, combined with lung ventilation images, we can evaluate the pulmonary shunt, dead space, V/Q ratio, to better clarify the physiological and pathological status of lung.This study intends to use EIT to evaluate pulmonary ventilation, blood flow distribution and local V/Q ratio before and after PPV, as well as to monitor the changes in pulmonary physiology before and after PPV, explore the mechanism of PPV improving oxygenation by combined with the changes in oxygenation, and explore the factors that predict and affect PPV responsiveness.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age ≥18 years. 2. Patients diagnosed with ARDS according to the Berlin definition and need to endotracheal intubated and mechanical ventilated in prone position within 48 hours of endotracheal intubation 3. PaO2/FiO2 < 150 mmHg with positive end-expiratory pressure (PEEP) ≥ 5 cmH2O according to the Berlin definition.

Exclusion Criteria:

* 1. Contraindications of EIT such as chest wound dressing, installation of pacemaker, defibrillator, etc.

  2. Unstable vertebral fracture 3. Within 15 days after severe facial trauma or facial surgery 4 within 15 days after tracheal surgery or sternotomy 5. Hemodynamic instability or recent cardiac arrest 6. Increased intraocular pressure. 7. Unstable femoral or pelvic fractures and pelvic external fixation. 8 He had severe chest wall disease and unstable rib fractures. 9 Recent cardiothoracic surgery. 10. Pneumothorax 11. Chronic lung disease: severe obstructive pulmonary disease, severe asthma, interstitial lung disease.

  12. Maternal 13. Extracorporeal membrane oxygenation(ECMO) had been administered on admission to the ICU.

  14. Intracranial hypertension 15. Pulmonary embolism, acute or chronic right heart failure 16. Severe cardiac dysfunction (New York Heart Association class III or IV, acute coronary syndrome, or sustained ventricular tachyarrhythmia), cardiogenic shock; 17. No informed consent was obtained

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who met inclusion exclusion criteria will implement EIT monitoring at the time of before the prone position, prone position for 16 hours and prone position ending 8h.
Sampling Method: Non-Probability Sample
Enrollment: 94 (Actual)
Dates: Start 2023-12-30 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2025-07-01 (Actual)

PRIMARY OUTCOMES:
Pulmonary ventilation perfusion(V/Q) ratio after 16 hours of PPV monitored by EIT | 16 hours after prone position ventilation
  the V/Q radio were monitored by EIT after patients were implemented prone position ventilation(PPV) for 16h. The images of ventilation distribution were collected by EIT, and the images of perfusion distribution were collected by injected 10ml of 10% hypertonic saline through a central vein catheter during inspiratory hold or expiratory hold. The ventilation and perfusion images were analysed by specialized software to obtain the data of V/Q radio.

SECONDARY OUTCOMES:
Pulmonary ventilation perfusion(V/Q) ratio before PPV monitored by EIT before PPV | within 1 hour before preparing PPV
  The V/Q radio were monitored by EIT before patients were implemented prone position ventilation(PPV). The images of ventilation distribution were collected by EIT, and the data of perfusion distribution were collected by injected 10ml of 10% hypertonic saline through a central vein catheter during inspiratory hold or expiratory hold. The ventilation and perfusion images were analysed by specialized software to obtain the data of V/Q radio.
Pulmonary ventilation perfusion(V/Q) ratio after PPV ending 8h monitored by EIT | 8 hours hours after prone position ventilation ending
  the V/Q radio were monitored by EIT 8 hours after prone position ventilation ending.The images of ventilation distribution were collected by EIT, and the data of perfusion distribution were collected by injected 10ml of 10% hypertonic saline through a central vein catheter during inspiratory hold or expiratory hold. The ventilation and perfusion images were analysed by specialized software to obtain the data of V/Q radio.
Pulmonary ventilation distribution before PPV, PPV for 16h and 8h after PPV ending | within 1hour before preparing PPV, 16 hours after and 8 hours after PPV ending
  Pulmonary ventilation distribution were monitored by EIT before PPV, PPV for 16h and 8h after PPV ending. The images of ventilation distribution were collected by EIT and analysed by specialized software to obtain the data.
Pulmonary perfusion distribution before PPV, PPV for 16h and 8h after PPV ending | within 1 hour before preparing PPV, 16 hours after and 8 hours after PPV ending
  The pulmonary perfusion distribution were monitored by EIT before PPV, PPV for 16h and 8h after PPV ending. The images of perfusion distribution were collected by injected 10ml of 10% hypertonic saline through a central vein catheter during inspiratory hold or expiratory hold. The perfusion images were analysed by specialized software to obtain the data of pulmonary perfusion distribution.
Pulmonary shunt percentage before PPV, PPV for 16h and 8h after PPV ending | within 1 hour before preparing PPV, 16 hours after and 8 hours after PPV ending
  The ventilation and perfusion images were analysed by specialized software to obtain the data of pulmonary shunt percentage.
Pulmonary dead space percentage before PPV, PPV for 16h and 8h after PPV ending | within 1 hour before preparing PPV, 16 hours after and 8 hours after PPV ending
  The ventilation and perfusion images were analysed by specialized software to obtain the data of pulmonary dead space percentage.
Peak pressure before PPV, PPV for 16h and 8h after PPV ending | Within 1 hour before preparing PPV, 16 hours after and 8 hours after PPV ending
  Peak pressure data were obtained from ventilators
Plat pressure before PPV, PPV for 16h and 8h after PPV ending | Within 1 hour before preparing PPV, 16 hours after and 8 hours after PPV ending
  Plat pressure data were obtained from ventilators
Tidal volume before PPV, PPV for 16h and 8h after PPV ending | within 1 hour before preparing PPV, 16 hours after and 8 hours after PPV ending
  Tidal volume data were obtained from ventilators
Driving pressure before PPV, PPV for 16h and 8h after PPV ending | within 1 hour before preparing PPV, 16 hours after and 8 hours after PPV ending
  Driving pressure(DP) data were obtained from ventilators
Static compliance(Cs) before PPV, PPV for 16h and 8h after PPV ending | within 1 hour before preparing PPV, 16 hours after and 8 hours after PPV ending
  Cs is equal to tidal volume divided by DP
P/F ratio before PPV, PPV for 16h and 8h after PPV ending | within 1 hour before preparing PPV, 16 hours after and 8 hours after PPV ending
  P/F ratio data were obtain from arterial blood gas analysis
Carbon dioxide partial pressure(PaCO2) before PPV, PPV for 16h and 8h after PPV ending | within 1 hour before preparing PPV, 16 hours after and 8 hours after PPV ending
  PaCO2 data were obtain from arterial blood gas analysis
Ventilatory ratio(VR) before PPV, PPV for 16h and 8h after PPV ending | within 1 hour before preparing PPV, 16 hours after and 8 hours after PPV ending
  VR=[minute ventilation (ml/min)×arterial partial tension of carbon dioxide (mmHg)] / [predicted body weight×100×37.5
28 days mortality | From the day of enrollment to day 28
  Mortality of from the day of enrollment to day 28
Ventilator free days(VFD) within 28 days | From the day of enrollment to day 28
  The number of ventilator free days for patients from enrollment day to day 28, if patients died within 28 days,VFD was equal to zero.
Mortality in the ICU | From the day of enrollment to the day of transfer from the ICU or death，up to 90 days
  Mortality in the ICU of all participants
Length of stay(LOS) | From the day of to the day of admitting to hospital to depart from the hospital or death，up to 90 days
  LOS(length of stay) of hospital

CONTACTS AND LOCATIONS:
Overall Officials: Xiaojing zou, MD, Principal Investigator — Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Locations (1):
- Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China

REFERENCES:
- [Background] Fan E, Brodie D, Slutsky AS. Acute Respiratory Distress Syndrome: Advances in Diagnosis and Treatment. JAMA. 2018 Feb 20;319(7):698-710. doi: 10.1001/jama.2017.21907. PMID 29466596
- [Background] Gierhardt M, Pak O, Walmrath D, Seeger W, Grimminger F, Ghofrani HA, Weissmann N, Hecker M, Sommer N. Impairment of hypoxic pulmonary vasoconstriction in acute respiratory distress syndrome. Eur Respir Rev. 2021 Sep 15;30(161):210059. doi: 10.1183/16000617.0059-2021. Print 2021 Sep 30. PMID 34526314
- [Background] Guerin C, Albert RK, Beitler J, Gattinoni L, Jaber S, Marini JJ, Munshi L, Papazian L, Pesenti A, Vieillard-Baron A, Mancebo J. Prone position in ARDS patients: why, when, how and for whom. Intensive Care Med. 2020 Dec;46(12):2385-2396. doi: 10.1007/s00134-020-06306-w. Epub 2020 Nov 10. PMID 33169218
- [Background] Guerin C, Reignier J, Richard JC, Beuret P, Gacouin A, Boulain T, Mercier E, Badet M, Mercat A, Baudin O, Clavel M, Chatellier D, Jaber S, Rosselli S, Mancebo J, Sirodot M, Hilbert G, Bengler C, Richecoeur J, Gainnier M, Bayle F, Bourdin G, Leray V, Girard R, Baboi L, Ayzac L; PROSEVA Study Group. Prone positioning in severe acute respiratory distress syndrome. N Engl J Med. 2013 Jun 6;368(23):2159-68. doi: 10.1056/NEJMoa1214103. Epub 2013 May 20. PMID 23688302
- [Background] Kharat A, Simon M, Guerin C. Prone position in COVID 19-associated acute respiratory failure. Curr Opin Crit Care. 2022 Feb 1;28(1):57-65. doi: 10.1097/MCC.0000000000000900. PMID 34750322
- [Background] Scaramuzzo G, Gamberini L, Tonetti T, Zani G, Ottaviani I, Mazzoli CA, Capozzi C, Giampalma E, Bacchi Reggiani ML, Bertellini E, Castelli A, Cavalli I, Colombo D, Crimaldi F, Damiani F, Fusari M, Gamberini E, Gordini G, Laici C, Lanza MC, Leo M, Marudi A, Nardi G, Papa R, Potalivo A, Russo E, Taddei S, Consales G, Cappellini I, Ranieri VM, Volta CA, Guerin C, Spadaro S; ICU-RER COVID-19 Collaboration. Sustained oxygenation improvement after first prone positioning is associated with liberation from mechanical ventilation and mortality in critically ill COVID-19 patients: a cohort study. Ann Intensive Care. 2021 Apr 26;11(1):63. doi: 10.1186/s13613-021-00853-1. PMID 33900484
- [Background] Lee HY, Cho J, Kwak N, Choi SM, Lee J, Park YS, Lee CH, Yoo CG, Kim YW, Lee SM. Improved Oxygenation After Prone Positioning May Be a Predictor of Survival in Patients With Acute Respiratory Distress Syndrome. Crit Care Med. 2020 Dec;48(12):1729-1736. doi: 10.1097/CCM.0000000000004611. PMID 33003079
- [Background] Clarke J, Geoghegan P, McEvoy N, Boylan M, Ni Choileain O, Mulligan M, Hogan G, Keogh A, McElvaney OJ, McElvaney OF, Bourke J, McNicholas B, Laffey JG, McElvaney NG, Curley GF. Prone positioning improves oxygenation and lung recruitment in patients with SARS-CoV-2 acute respiratory distress syndrome; a single centre cohort study of 20 consecutive patients. BMC Res Notes. 2021 Jan 9;14(1):20. doi: 10.1186/s13104-020-05426-2. PMID 33422143
- [Background] Bachmann MC, Morais C, Bugedo G, Bruhn A, Morales A, Borges JB, Costa E, Retamal J. Electrical impedance tomography in acute respiratory distress syndrome. Crit Care. 2018 Oct 25;22(1):263. doi: 10.1186/s13054-018-2195-6. PMID 30360753
- [Background] Wang YX, Zhong M, Dong MH, Song JQ, Zheng YJ, Wu W, Tao JL, Zhu L, Zheng X. Prone positioning improves ventilation-perfusion matching assessed by electrical impedance tomography in patients with ARDS: a prospective physiological study. Crit Care. 2022 May 27;26(1):154. doi: 10.1186/s13054-022-04021-0. PMID 35624489
- [Background] Fan E, Del Sorbo L, Goligher EC, Hodgson CL, Munshi L, Walkey AJ, Adhikari NKJ, Amato MBP, Branson R, Brower RG, Ferguson ND, Gajic O, Gattinoni L, Hess D, Mancebo J, Meade MO, McAuley DF, Pesenti A, Ranieri VM, Rubenfeld GD, Rubin E, Seckel M, Slutsky AS, Talmor D, Thompson BT, Wunsch H, Uleryk E, Brozek J, Brochard LJ; American Thoracic Society, European Society of Intensive Care Medicine, and Society of Critical Care Medicine. An Official American Thoracic Society/European Society of Intensive Care Medicine/Society of Critical Care Medicine Clinical Practice Guideline: Mechanical Ventilation in Adult Patients with Acute Respiratory Distress Syndrome. Am J Respir Crit Care Med. 2017 May 1;195(9):1253-1263. doi: 10.1164/rccm.201703-0548ST. PMID 28459336
- [Background] Bellani G, Laffey JG, Pham T, Fan E, Brochard L, Esteban A, Gattinoni L, van Haren F, Larsson A, McAuley DF, Ranieri M, Rubenfeld G, Thompson BT, Wrigge H, Slutsky AS, Pesenti A; LUNG SAFE Investigators; ESICM Trials Group. Epidemiology, Patterns of Care, and Mortality for Patients With Acute Respiratory Distress Syndrome in Intensive Care Units in 50 Countries. JAMA. 2016 Feb 23;315(8):788-800. doi: 10.1001/jama.2016.0291. PMID 26903337
- [Background] Langer T, Brioni M, Guzzardella A, Carlesso E, Cabrini L, Castelli G, Dalla Corte F, De Robertis E, Favarato M, Forastieri A, Forlini C, Girardis M, Grieco DL, Mirabella L, Noseda V, Previtali P, Protti A, Rona R, Tardini F, Tonetti T, Zannoni F, Antonelli M, Foti G, Ranieri M, Pesenti A, Fumagalli R, Grasselli G; PRONA-COVID Group. Prone position in intubated, mechanically ventilated patients with COVID-19: a multi-centric study of more than 1000 patients. Crit Care. 2021 Apr 6;25(1):128. doi: 10.1186/s13054-021-03552-2. PMID 33823862